CLINICAL TRIAL: NCT02670993
Title: Support by Singing Sessions on Physical and Moral Pain : Assessment of Its Effectiveness in Alzheimer's Disease. Multicenter Study LACME
Brief Title: Support by Singing Sessions on Physical and Moral Pain : Assessment of Its Effectiveness in Alzheimer's Disease
Acronym: LACME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1508071; 2015-A01404-45 (Other: ANSM)
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group : Singing sessions. (Experimental): Patients will participate to singing working sessions. They will continue to take their usual treatments during the study period.
  Interventions: Behavioral: Singing sessions.
- Control group : Painting sessions. (Active Comparator): Patients will continue to participate to painting work sessions, and to take their usual treatments during the study.
  Interventions: Behavioral: Painting sessions.

INTERVENTIONS:
Behavioral: Singing sessions. — Patients will be in singing work groups, and will participate to these sessions during 12 weeks, with one session per week of 2 hours.
  Arms: Control group : Singing sessions.
Behavioral: Painting sessions. — Patients will be in painting groups, they will participate to this work session during 12 weeks, with one session of 2 hours per week.
  Arms: Control group : Painting sessions.

SUMMARY:
Alzheimer Disease (AD), characterized by cognitive and psycho-behavioral troubles, concerns essentially 65 years old and older patients. Antalgic and psychotropic treatments have adverse effects in old people, and have to be used carefully. To improve the pain support and limit the drug consumption, it is possible to perform therapies without drugs. Among them, musical intervention represents an interesting complementary support, to deal with physical and moral pain in AD.

DETAILED DESCRIPTION:
Alzheimer Disease (AD), characterized by cognitive and psycho-behavioral troubles, concerns essentially 65 years old and older patients. At this age, comorbidities are frequent and numerous, and often linked to pain. The prevalence is comprised between 40 and 85% according to different studies. Antalgic and psychotropic treatments have adverse effects in old people, and have to be used carefully. To improve the pain support and limit the drug consumption, it is possible to perform therapies without drugs. Among them, musical intervention represents an interesting complementary support, to deal with physical and moral pain in AD.

The primary outcome is to evaluate the singing support on physical pain, by comparison with a control activity : "painting session".

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years old and older, fulfilling the diagnostic criteria for Alzheimer's disease to a mild dementia stage, or mild cognitive impairment
* Delay of at least one month between the diagnosis and the early work sessions
* If use of psychotropic drugs, they must be stabilized for 3 month
* If analgesics consumption level 2 or 3 they must be stabilized for 1 month
* With a score greater than or equal to 22 on the simplified visual scale (EVS) pain.
* Visual capabilities , auditory and oral or written expression in French language sufficient for conducting clinical and neuropsychological evaluations;
* MMSE > 20
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Patient with a different etiology of cognitive disorder that of Alzheimer's disease
* Patients with severe disease, progressive or unstable nature which may interfere with the evaluation variables
* Patient with blindness or deafness could compromise its assessment
* Patient under guardianship

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Score at the EVS = simplified visual scale | Month 1
  To evaluate the efficacy of the singing sessions on pain in Alzheimer's Disease patients (beginning stage), by comparison with a control activity (painting), on pain intensity.

SECONDARY OUTCOMES:
Score at the EN (digital scale) scale | Month 1
  To evaluate the efficacy of the singing sessions on pain in Alzheimer's Disease patients (beginning stage), by comparison with a control activity (painting), on pain intensity.
Score at the BPI (Brief Pain Inventory) scale : Brief pain Inventory | Month 1
  To evaluate the efficacy of the singing sessions on pain in Alzheimer's Disease patients (beginning stage), by comparison with a control activity (painting), on pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: ROUCH Isabelle, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Hospices civils de Lyon, Lyon
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No